CLINICAL TRIAL: NCT00017693
Title: Phase II Efficacy Study of Aerosolized Recombinant Human IL-4 Receptor in Asthma
Brief Title: Recombinant Human IL-4 Receptor Used in Treatment of Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT Asthma 013.0014; NCT00016705 (obsolete NCT alias)
Record Dates: First submitted 2001-06-07; First posted 2001-08-31 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: Recombinant Proteins; Aerosols; Asthma; Receptors, Interleukin-4; Forced Expiratory Volume
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 0.75mg rsIL-4R (Experimental): Recombinant human soluble IL-4 receptor (rsIL-4R) given by means of inhalation once weekly for 12 weeks. The study drug was administered in the clinic at a final volume of 2.5 mL in sterile normal saline solution with a breath-assisted Pari LC Star nebulizer powered by a Proneb Turbo portable compressor.
  Interventions: Biological: Recombinant human soluble IL-4 receptor
- 1.5mg rsIL-4R (Experimental): Recombinant human soluble IL-4 receptor (rsIL-4R) given by means of inhalation once weekly for 12 weeks. The study drug was administered in the clinic at a final volume of 2.5 mL in sterile normal saline solution with a breath-assisted Pari LC Star nebulizer powered by a Proneb Turbo portable compressor.
  Interventions: Biological: Recombinant human soluble IL-4 receptor
- 3.0mg rsIL-4R (Experimental): Recombinant human soluble IL-4 receptor (rsIL-4R) given by means of inhalation once weekly for 12 weeks. The study drug was administered in the clinic at a final volume of 2.5 mL in sterile normal saline solution with a breath-assisted Pari LC Star nebulizer powered by a Proneb Turbo portable compressor.
  Interventions: Biological: Recombinant human soluble IL-4 receptor
- Placebo for rsIL-4R (Placebo Comparator): The placebo for recombinant human soluble IL-4 receptor (rsIL-4R) consisted of identically prepared excipient in the same volume (2.5 mL). To maintain blinding, medication was dispensed by an individual who was not responsible for patient care or assessment. Treatment assignment was blinded to all personnel involved in direct conduct or monitoring of the study.
  Interventions: Biological: Placebo for Recombinant human soluble IL-4 receptor

INTERVENTIONS:
Biological: Recombinant human soluble IL-4 receptor — Subjects were randomized to twelve once weekly nebulizations of 0.75, 1.5, or 3.0 mg dose of recombinant human soluble IL-4 receptor (rsIL-4R)
  Arms: 0.75mg rsIL-4R; 1.5mg rsIL-4R; 3.0mg rsIL-4R
Biological: Placebo for Recombinant human soluble IL-4 receptor — Subjects were randomized to twelve once weekly nebulizations of placebo for recombinant human soluble IL-4 receptor (rsIL-4R). Identically prepared (to the recombinant human soluble IL-4 receptor) in the same volume
  Other Names: Placebo Treatment
  Arms: Placebo for rsIL-4R

SUMMARY:
The purpose is to measure the effectiveness of recombinant human interleukin-4 receptor (IL-4R) in treating asthma.

Asthma can be caused by the allergic response from breathing in certain irritants. Interleukin 4 (IL-4), which is naturally produced by the body, plays a major role in this allergic response. Doctors feel that IL-4 activity may be stopped by giving IL-4R, a product that binds to IL-4, and thereby decrease the problems of asthma.

DETAILED DESCRIPTION:
A major factor in the pathogenesis of asthma is the development of an allergic inflammatory response to inhaled antigens. Interleukin-4 (IL-4) plays a key role in this response. Binding and inactivating the IL-4 molecule with IL-4R may diminish the allergic asthmatic response by inhibiting activities of IL-4.

Patients are randomized to 1 of 3 treatment groups and, within each group, are stratified by baseline FEV1 cohort. Patients receive either dose level 1 of IL-4R, dose level 2 of IL-4R, or placebo, by aerosol drug delivery device, once a week for 12 weeks. There are frequent clinic visits and several follow-up visits. Physical exams and spirometry are done regularly; immunizations are administered on Day 28; and a skin tests panel is given on Day 84. Blood samples are collected at study visits during treatment and follow-up to test for immunology/serology parameters, chemistry profiles, and asthma-related DNA polymorphisms. Patients are provided with peak flow meters and must demonstrate their proper use so that a peak expiratory flow (PEF) diary and a symptoms diary can be maintained. Selected sites measure exhaled nitric oxide and collect induced sputum samples. Assessments for adverse events are conducted at 16 and 40 weeks following the first study drug treatment.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 12 to 85 years of age (consent of parent or guardian required if under 18 years).
* Have continuous asthma and are being treated with albuterol MDI only.
* Have reduced lung functions.
* Have a positive reaction to 2 substances as demonstrated with a skin test.
* Have been a nonsmoker for at least 2 years and have not smoked more than 1 pack a day for 5 years or less.
* Agree to use contraception throughout the study.
* Agree not to donate blood throughout the study.
* Are able to use correctly an aerosol drug delivery device.
* Have had an asthma attack on at least 3 of the last 7 days.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Had asthma requiring hospitalization within 6 weeks of beginning study treatment.
* Had asthma requiring emergency room treatment within 12 months of beginning study treatment.
* Had a respiratory infection that affected asthma within 2 weeks of beginning study treatment.
* Had a breathing tube inserted for asthma treatment within 15 years of beginning study treatment.
* Were previously enrolled in a study of soluble IL-4 receptor.
* Have drug abuse, alcohol abuse, or a mental illness that may interfere with the study.
* Have serious medical problems (such as heart or lung problems, uncontrolled high blood pressure, are overweight to the extent that ability to breathe is affected, or have cancer other than skin cancer), diabetes, autoimmune diseases, or HIV.
* Are pregnant or breast-feeding.
* Have used certain drugs.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 1998-05; Primary Completion 2000-02 (Actual); Study Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Forced expiratory volume in 1 second (FEV1) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Larry Borish, MD, Study Chair — University of Virginia; Harold Nelson, MD, Study Chair — National Jewish Health

REFERENCES:
- [Result] Borish LC, Nelson HS, Corren J, Bensch G, Busse WW, Whitmore JB, Agosti JM; IL-4R Asthma Study Group. Efficacy of soluble IL-4 receptor for the treatment of adults with asthma. J Allergy Clin Immunol. 2001 Jun;107(6):963-70. doi: 10.1067/mai.2001.115624. PMID 11398072
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/